CLINICAL TRIAL: NCT00580814
Title: Brain Dopamine Function in Adults With ADHD
Acronym: Brookhaven
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Duke University (Other)
Responsible Party: Principal Investigator, Coleen Cunningham, Professor and Chair of Pediatrics, University of California, Irvine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20054659
Record Dates: First submitted 2007-10-04; First posted 2007-12-27 (Estimated); Results first posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Brookhaven; ADHD; Dopamine; methylphenidate; PET
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylphenidate (Experimental): intervention is methylphenidate once daily for 12 months, doses individually titrated
  Interventions: Drug: Experimental: methylphenidate treatment
- No medication (No Intervention): no methylphenidate treatment for non ADHD

INTERVENTIONS:
Drug: Experimental: methylphenidate treatment — subjects received mehtylphenidate treatment for 12 months
  Other Names: methylphenidate once daily for 12 months, doses individually titrated for efficacy
  Arms: methylphenidate

SUMMARY:
The purpose of the study is to investigate the functional state of dopamine cells and the dopamine transporter in ADHD subjects and controls to assess the effects of chronic methylphenidate treatment on dopamine cell function and dopamine transporter levels in ADHD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must give informed consent
* Must be between the ages of 18 and 45 years old.
* Must have a confirmed diagnosis of ADHD
* Must have scored on a rating scale that indicate a significant level of symptom severity.
* Must have a childhood history of ADHD must be documented using established test criteria.
* Must have had no previous medication treatment for ADHD except for a short term treatment period of less than three months, which should have occurred at least six months prior to the study.
* Must have an interest in receiving long-term medication treatment for ADHD.

Exclusion Criteria:

* Must not test positive for psychoactive drugs during a urine drug screen.
* Must not be pregnant.
* Must not be breastfeeding.
* Must have no past or present history of dependence on alcohol or other drugs of abuse except nicotine or caffeine.
* Must have no past or present history of a psychiatric disorder except ADHD.
* Must have no medical illness that may affect brain function.
* Must not have taken medication that may affect brain function.
* Must not have had head trauma with loss of consciousness (> 30 minutes).
* Must not have significant anxiety or depression as determined by an established test.
* Must have no history of a significant learning disability.
* Must have no history of cardiovascular or endocrinological disease.
* Must have no history of coagulation disorder.
* Must have no history of sensitivity to lidocaine and/or prilocaine.
* Must have no history of claustrophobia.
* Contraindication to MRI environment (presence of any implanted metallic objects such as cardiac/neural pacemakers, defibrillators, aneurysm clips, certain heart valves, spinal nerve stimulators, artificial joints/limbs, shrapnel/bullets, metal fragments in their eyes, cochlear implants, hearing aids, dental implants).
* Must have no history of glaucoma.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-02; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Wigal, Ph.D., Principal Investigator — UC Irvine
Locations (1):
- UCI Child Development Center, Irvine, California, United States

REFERENCES:
- [Background] Wang GJ, Volkow ND, Wigal T, Kollins SH, Newcorn JH, Telang F, Logan J, Jayne M, Wong CT, Han H, Fowler JS, Zhu W, Swanson JM. Long-term stimulant treatment affects brain dopamine transporter level in patients with attention deficit hyperactive disorder. PLoS One. 2013 May 15;8(5):e63023. doi: 10.1371/journal.pone.0063023. Print 2013. PMID 23696790
- [Result] Volkow, N.d., Wand, G., Kollins., Wigal, T., Newcorn, J., Telang, F., Fowler, J., Solanto, M.V., Logan, J., Ma, Y., Pradham. K., Wong, C., Zhu, W. & Swanson, J.M. Dopamine Reward Pathway Disrupted in Patients with ADHD: Therapeutic Implications, Journal of American Medical Association.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 3 sites from 2004 - 2008. They were all consented to the protocol before any study procedures were done.Subjects were recruited through flyers and newspaper ads. They were seen at medical clinics and ADHD diagnosis was confirmed. All subjects were treatment naive for stimulant medications.
Pre-assignment Details: Subjects were interviewed to determine mental health diagnosis of ADHD with symptoms existing since childhood. All other psychiatric diagnoses were exclusionary as was neurological or cerebral disease. Healthy controls were also recruited. All subjects were then scheduled for scans at Brookhaven and ADHD subjects then recieved one year of meds.
Groups:
- Methylphenidate Treatment: methylphenidate treatment
  methylphenidate : Subjects (18) in this arm recieved methylphenidate for one year.
- no Intervention: no intervention for 12 months
  no intervention : no treatment for 11 subjects for 12 months
Period: Baseline PET Scans at Brookhaven
Arm/Group | Methylphenidate Treatment | no Intervention
Started | 55 | 20
Completed | 55 | 20
Not Completed | 0 | 0
Period: One Year of Treatment or no Intervention
Arm/Group | Methylphenidate Treatment | no Intervention
Started | 55 | 20
Completed | 18 | 11
Not Completed | 37 | 9
Period: Repeated PET Scans
Arm/Group | Methylphenidate Treatment | no Intervention
Started | 18 | 11
Completed | 18 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methylphenidate Treatment | no Intervention | Total
Number analyzed (Participants) | 55 | 20 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 55 | 20 | 75
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (1.9) | 33.2 (1.6) | 31.5 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 12 | 42
  Male | 25 | 8 | 33
Region of Enrollment [Number; unit: participants]
  United States | 55 | 20 | 75
PET scan of DAT availability [Number; unit: participants] — All subjects who are enrolled will receive PET scans at Brookhaven to examine DAT availability
  participants | 55 | 20 | 75

OUTCOME MEASURES:

1. Primary Outcome: DAT Availability
Description: Striatal DAT availability as noted in PET scans post one year of methylphenidate treatment or no intervention.
  The unit listed as binding potential (BPND) was measured with a dynamic PET scan protocol, using carbon-11 labeled cocaine, a radioligand with specific binding to DAT (which is inhibited by drugs that block DAT but not by drugs that block the norephephrine or serotonin transporters). This radiotracer was utilized to quantify DAT availability as non-displaceable binding potential using a standard kinetic model for reversible ligands.
  The dynamic PET scans were started immediately after injection of [11C]cocaine (specific activity 0.5-1.5 Ci/uM at end of bombardment). Arterial blood was obtained to measure the concentration of unchanged [11C] cocaine in plasma for quantification of DAT availability.
Time Frame: 1 year
Population: DAT availability was measured as ratio of distribution volume in striatum to cerebellum -1 (BPND-1), which represents number of transporters free to bind radiotracer. Distribution volume ratio images were transformed into images by computing total distribution volume in each pixel and dividing by distribution volume in cerebellum. Regions of interest in striatum (caudate, putamen, ventral striatum) were drawn on an averaged emission image (10 to 60 minutes for [11C] cocaine).
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Methylphenidate Treatment | no Intervention
Number analyzed (Participants) | 18 | 11
ratio | 2.68 (0.28) | 2.85 (0.31)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Subjects seen monthly for one year.
Arm/Group | Methylphenidate Treatment | no Intervention
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/20
Other Adverse Events (participants affected / at risk) | 0/55 | 0/20

LIMITATIONS AND CAVEATS:
The length of the study resulted in the loss of a number of subjects in both arms of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No